CLINICAL TRIAL: NCT03227302
Title: Associations of the Grades of Doctor and Neonatal Outcomes: An Observational Prospective Study
Brief Title: Associations of the Grades of Doctor and Neonatal Outcomes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Responsible Party: Principal Investigator, Ma Juan, Principal Investigator, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Other Study IDs: grades of doctor and neonaltal
Record Dates: First submitted 2017-06-30; First posted 2017-07-24 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Standardized Training System for Residents; Neonatal Outcomes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- attending obstetrician: the low grade doctor who can do caesarean operation with no pregnant complications.
  Interventions: Procedure: attending obstetrician
- associate chief obstetrician: The middle grade doctor who can do caesarean operation with no or mild or middle pregnant complications.
  Interventions: Procedure: associate obstetrician
- chief obstetrician: the high doctor who can do all caesarean operation without limitations
  Interventions: Procedure: chief obstetrician

INTERVENTIONS:
Procedure: attending obstetrician — Attending obstetrician can do the caesarean operation without pregnant complications.
  Groups: attending obstetrician
Procedure: associate obstetrician — Associate chief Obstetrician can do the caesarean operation without or mild or middle pregnant complications.
  Groups: associate chief obstetrician
Procedure: chief obstetrician — Chief obstetrician can do all caesarean operation without limitations.
  Groups: chief obstetrician

SUMMARY:
In China, the standardized training system for residents was built last year, and the associations of the grades of doctors and accoucheurs and neonatal outcomes remains unclear.

DETAILED DESCRIPTION:
In China, the grades of doctors and accoucheurs are divided into four levels, and different levels may induce differences of neonatal asphyxia and death. The standardized training system for residents was built last year,the associations of the grades of doctors and accoucheurs and neonatal asphyxia,neonatal death before and after the training systems need to be assess.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age (GA) is from 26 to 42 weeks

Exclusion Criteria:

* major congenital malformations or complex congenital heart disease

Ages: 1 Minute to 100 Days | Sex: All
Age Groups: Child
Study Population: All neonates with gestational age are from 26 weeks to 42 weeks
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
neonatal asphyxia | within 28 days
  neonatal asphyxia was defined according to manual of neonatal care
death | within 28 days
  neonatal death

SECONDARY OUTCOMES:
Bayley Scales of Infant Development | at 2 months and 2 years old
  to assess the development using Bayley Scales of Infant Development

CONTACTS AND LOCATIONS:
Overall Officials: Shi Yuan, PhD,MD, Study Director — Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Locations (1):
- Department of Pediatrics, Daping Hospital, Third Military Medical University, Chongqing, Chongqing Municipality, China